CLINICAL TRIAL: NCT02157051
Title: A Phase I Trial of the Safety and Immunogenicity of a Multiple Antigen Vaccine (STEMVAC) in HER2 Negative Advanced Stage Breast Cancer Patients
Brief Title: Vaccine Therapy in Treating Patients With HER2-Negative Stage III-IV Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Breast Cancer Alliance (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 9140; NCI-2014-01070 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 137; 9140 (Other: Fred Hutch/University of Washington Cancer Consortium); RG1715017 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2014-06-03; First posted 2014-06-05 (Estimated); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: HER2 Negative Breast Carcinoma; Recurrent Breast Carcinoma; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer; Stage III Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (STEMVAC) (Experimental): Patients receive CD105/Yb-1/SOX2/CDH3/MDM2-polyepitope plasmid DNA vaccine with rhuGM-CSF as 1 injection ID every 28 days for 3 months. Patients may also receive 2 additional booster STEMVAC vaccines at 3 and 9 months after the third vaccine in the absence of unacceptable toxicity or disease progression.
  Interventions: Biological: CD105/Yb-1/SOX2/CDH3/MDM2-polyepitope Plasmid DNA Vaccine; Other: Laboratory Biomarker Analysis
- Arm 2 (STEMVAC) (Experimental): Patients receive CD105/Yb-1/SOX2/CDH3/M2-polyepitope plasmid DNA vaccine with rhuGM-CSF as 2 injections ID every 28 days for 3 months. Patients may also receive 2 additional booster STEMVAC vaccines at 3 and 9 months after the third vaccine in the absence of unacceptable toxicity or disease progression.
  Interventions: Biological: CD105/Yb-1/SOX2/CDH3/MDM2-polyepitope Plasmid DNA Vaccine; Other: Laboratory Biomarker Analysis
- Arm 3 (STEMVAC) (Experimental): Patients receive CD105/Yb-1/SOX2/CDH3/MDM2-polyepitope plasmid DNA vaccine with rhuGM-CSF as 3 injections ID every 28 days for 3 months. Patients may also receive 2 additional booster STEMVAC vaccines at 3 and 9 months after the third vaccine in the absence of unacceptable toxicity or disease progression.
  Interventions: Biological: CD105/Yb-1/SOX2/CDH3/MDM2-polyepitope Plasmid DNA Vaccine; Other: Laboratory Biomarker Analysis
- Arm 4 (STEMVAC) (Experimental): Patients receive CD105/Yb-1/SOX2/CDH3/MDM2-polyepitope plasmid DNA vaccine with rhuGM-CSF as 2 injections ID every 28 days for 3 months. Patients may also receive 1 additional STEMVAC vaccine at 3 months after the third vaccine in the absence of unacceptable toxicity or disease progression.
  Interventions: Biological: CD105/Yb-1/SOX2/CDH3/MDM2-polyepitope Plasmid DNA Vaccine; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: CD105/Yb-1/SOX2/CDH3/MDM2-polyepitope Plasmid DNA Vaccine — Given ID
  Other Names: CD105/Yb-1/SOX2/CDH3/MDM2 Plasmid Vaccine; STEMVAC; STEMVAC Th1 Polyepitope Plasmid-based Vaccine
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of multiantigen deoxyribonucleic acid (DNA) plasmid-based vaccine in treating patients with human epidermal growth factor receptor 2 (HER2)-negative stage III-IV breast cancer. Multiantigen DNA plasmid-based vaccine may target immunogenic proteins expressed in breast cancer stem cells which are the component of breast cancer that is resistant to chemotherapy and has the ability to spread. Vaccines made from DNA may help the body build an effective immune response to kill tumor cells.

DETAILED DESCRIPTION:
OUTLINE: This is a dose-escalation study. Patients are assigned to 1 of 4 arms.

Arm 1: Patients receive CD105/Yb-1/SOX2/CDH3/MDM2-polyepitope plasmid DNA vaccine with recombinant human granulocyte-macrophage colony-stimulating factor (rhuGM-CSF) as 1 injection intradermally (ID) every 28 days for 3 months. Patients may also receive 2 additional booster STEMVAC vaccines at 3 and 9 months after the third vaccine in the absence of unacceptable toxicity or disease progression.

ARM 2: Patients receive CD105/Yb-1/SOX2/CDH3/M2-polyepitope plasmid DNA vaccine with rhuGM-CSF as 2 injections ID every 28 days for 3 months. Patients may also receive 2 additional booster STEMVAC vaccines at 3 and 9 months after the third vaccine in the absence of unacceptable toxicity or disease progression.

ARM 3: Patients receive CD105/Yb-1/SOX2/CDH3/MDM2-polyepitope plasmid DNA vaccine with rhuGM-CSF as 3 injections ID every 28 days for 3 months. Patients may also receive 2 additional booster STEMVAC vaccines at 3 and 9 months after the third vaccine in the absence of unacceptable toxicity or disease progression.

ARM 4: Patients receive CD105/Yb-1/SOX2/CDH3/MDM2-polyepitope plasmid DNA vaccine with rhuGM-CSF as 2 injections ID every 28 days for 3 months. Patients may also receive 1 additional STEMVAC vaccine at 3 months after the third vaccine in the absence of unacceptable toxicity or disease progression.

After completion of study treatment, patients are followed up twice yearly for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage III-IV HER2 negative breast cancer treated with primary or salvage therapy and now have:

  * No evidence of disease (NED), or
  * Stable bone only disease
* Patients who have completed standard of care and recovered with mild to no residual toxicity from recent therapy
* Patients must be at least 28 days post cytotoxic chemotherapy, and/or monoclonal antibody therapy (excluding bone-directed therapy), prior to enrollment
* Patients must be at least 28 days post systemic steroids prior to enrollment
* Patients on bisphosphonates, denosumab, and/or endocrine therapy are eligible
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status score of =< 1
* Patients must have recovered from major infections and/or surgical procedures, and in the opinion of the investigator, not have any significant active concurrent medical illnesses precluding protocol treatment
* Estimated life expectancy of more than 6 months
* White blood cells (WBC) >= 3000/mm^3 (within 30 days of first vaccination)
* Lymphocyte count >= 800/mm^3 (within 30 days of first vaccination)
* Platelet count >= 75,000/mm^3 (within 30 days of first vaccination)
* Hemoglobin (Hgb) >= 10 g/dl (within 30 days of first vaccination)
* Serum creatinine <= 1.2 mg/dl or creatinine clearance > 60 ml/min (within 30 days of first vaccination)
* Total bilirubin <= 1.5 mg/dl (within 30 days of first vaccination)
* Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) <= 2 times upper limit of normal (ULN) (within 30 days of first vaccination)
* Blood glucose < 1.5 ULN (within 30 days of first vaccination)
* All patients who are having sex that can lead to pregnancy must agree to contraception for the duration of study

Exclusion Criteria:

* Patients with any of the following cardiac conditions:

  * Symptomatic restrictive cardiomyopathy
  * Unstable angina within 4 months prior to enrollment
  * New York Heart Association functional class III-IV heart failure on active treatment
  * Symptomatic pericardial effusion
* Patients at risk for gastrointestinal bleeding (example: peptic ulcer disease, prolonged daily non-steroidal anti-inflammatory use)
* Patients with any seizure disorder
* Patients with any contraindication to receiving rhuGM-CSF based products
* Patients with any clinically significant autoimmune disease uncontrolled with treatment
* Patients who are simultaneously enrolled in any other treatment study
* Patients who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2027-02-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of toxicity per Cancer Therapy Evaluation Program Common Terminology Criteria for Adverse Events version 4.0 | Up to 1 month after last vaccine
  The type and grade of toxicities noted during the immunization regimen will be summarized. Adverse events noted by the investigator/designated clinical research staff will be tabulated according to the affected body system. Descriptive statistics will be used to summarize changes from baseline in clinical and/or laboratory parameters.
Immunologic efficacy defined as achievement of a statistically significant increase in Th1 cell immunity for at least 50% of the immunizing antigens as compared to baseline | Up to 5 years

SECONDARY OUTCOMES:
Memory Th1 dominant immune response to all five antigens over time | Up to 12 months
Modulation of T-regulatory (Treg) cells with vaccination | Up to 12 months
  Treg defined as present or absent, and the probability will be estimated as a simple proportion.
Modulation of MDSC with vaccination | Up to 12 months
  MDSC defined as present or absent, and the probability will be estimated as a simple proportion.
STEMVAC specific Type 1 immune response | Up to 12 months
  Will detect if STEMVAC specific Type 1 immune response would be negatively correlated with the type II bacterial-tumor antigen (Bac-TA) specific responses. Statistical strategies will be used to assess the incidence and breadth of vaccine induced immunity as related to the levels of Bac-TA Th2 (Arm 4). For magnitude, the initial analysis could include two-tailed Pearson's correlation or even two tailed T tests between clear responder and non-responders. Specific organisms in the gut microbiome may prevent the development of tumor specific Type I immunity after vaccination, and will be evaluated by flow cytometry of peripheral blood mononuclear cells. Analysis could identify a blood based biomarker (Bac-TA responses) that could identify patients who would be less responsive to immune modulation and will be assessed by shotgun metagenomic sequencing.
Bac-TA cross-reactive T-cells | Up to 12 months
  Will evaluate whether organisms associated with Bac-TA cross-reactive T-cells are represented in the patient's microbiome. Will be assessed by collecting stool with the OMNIgene-GUT collection Kits (DNA Genotek) (Arm 4). Analysis could identify a blood based biomarker (Bac-TA responses) that could identify patients who would be less responsive to immune modulation and will be assessed by shotgun metagenomic sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Disis, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No